CLINICAL TRIAL: NCT05155722
Title: A Phase I Dose Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerance and Pharmacokinetic of BAT1308 Injection in Patients With Advanced Solid Tumors
Brief Title: Assessment of Safety ,Tolerance and Pharmacokinetics Clinical Efficacy With BAT1308 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-1308-001-CR
Record Dates: First submitted 2021-11-18; First posted 2021-12-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): First Phase: dose escalation study. It was divided into three dose groups: 100mg, 300mg and 600mg. The safety, tolerance and pharmacokinetics of BAT1308 injection were explored according to the 3+3 dose increasing mode. It is expected that 12-18 cases will be included in the group. Second Phase: dose expansion study. After the completion of dose increment, 300mg tolerated doses were selected for extended research on advanced non-small cell lung cancer, advanced hepatocellular carcinoma and cervical cancer (80-130 cases), so as to provide recommended doses for subsequent clinical trials.
  Interventions: Drug: BAT1308

INTERVENTIONS:
Drug: BAT1308 — A 21 day treatment cycle was administered every 3 weeks (Q3W) on day 1 of each cycle. Six consecutive dosing cycles are recommended for the dose escalation phase. In the extended study phase, after the end of the 6th treatment cycle, after the risk and benefit are evaluated by the investigator in combination with the clinical practice, if the subjects are still in a state of clinical benefit (including CR, PR and SD), the investigator can decide to appropriately extend the treatment of BAT1308. Until disease progression, unacceptable toxicity, withdrawal of informed consent, loss of follow-up, death, acceptance of new antitumor therapy, termination of treatment by investigator evaluation, or 12 months after initial administration, whichever is the earliest.

SUMMARY:
A phase I dose escalation and cohort expansion study to evaluate the safety, tolerance and pharmacokinetic of BAT1308 injection in patients with advanced solid tumors

DETAILED DESCRIPTION:
This study is a multicenter, open, dose-increasing and dose-expanding phase I clinical study. The dose increasing method of "3 + 3" is used to explore the safety, tolerance and pharmacokinetic characteristics of BAT1308 injection in patients with advanced solid tumors (12-18 cases). After the completion of dose increment, 300mg tolerated doses were selected for extended research on advanced non-small cell lung cancer, advanced hepatocellular carcinoma and cervical cancer (80-130 cases), so as to provide recommended doses for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (including boundary value), male or female;
2. Voluntarily sign informed consent;
3. Research Population:

   A) Dose escalation stage: patients with advanced malignant solid tumors that have been pathologically confirmed, failed or are intolerant to standard therapy. Agree to provide previously stored tumor tissue samples for PD-L1 testing or existing PD-L1 testing results.

   B) Dose extension phase: divided into 3 cohorts:

   i. Cohort A: pathologically confirmed patients with advanced non-small cell lung cancer (NSCLC) who failed standard therapy and who were intolerant or refused standard therapy. And agree to provide previously stored tumor tissue specimens or fresh biopsy of tumor focal tissue for relevant pathological test pD-L1 ≥1% or existing test results show PD-L1≥1%, ii. Cohort B: Patients with advanced hepatocellular carcinoma (HCC) confirmed by pathological or clinical diagnosis, who failed standard therapy, were intolerant or refused standard therapy, had no PD-L1 test requirements, had child-Pugh liver function rating of GRADE A and better grade B (≤7 points), and had no history of hepatic encephalopathy.

   iii. Queue C: through pathology diagnosed with cervical cancer (pathological type squamous carcinoma or gland scale cancer), the phase of recurrence or metastasis (2018 edition FIGO stage IVB), cervical cancer, the stage of recurrence or metastasis after standard treatment (first-line platinum-based chemotherapy medicine + beacizumab bead sheet resistance treatment) after failure, intolerance, or refused to accept the standard treatment for patients. Agree to provide previously stored tumor tissue samples or fresh biopsy of tumor focus tissue (exemption if no previously stored tumor tissue samples are available and the investigator assesses there is a significant risk of reacquisition).
4. According to recist1.1 standard, there is at least one measurable tumor focus;
5. ECOG score shall be 0 or 1;
6. The investigator assessed the expected survival ≥ 12 weeks;
7. Have sufficient organ and bone marrow functions as below:Blood routine (no blood transfusion, no hematopoietic stimulator, and no medication to correct blood count within 14 days prior to first dosing),Neutrophil absolute count (ANC) ≥1.5 x 109 /L, Platelet count ≥75×109/L, Hemoglobin≥9g/dL 或≥5.6mmol/L, Blood coagulation function Prothrombin time (PT) or International standardized ratio (INR) and activated partial thrombin time (APTT) ≤ 1.5×ULN, Liver function Total bilirubin (TBIL) ≤2×ULN ,Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤3×ULN(Other solid tumors without liver metastasis) or ≤5×ULN (Hepatocellular carcinoma, or liver metastases), Serum Creatinine ≤1.5×ULN ，renal function Serum creatinine clearance rate>60ml/min (Cockcroft-Gault formula), Thyroid function: Abnormalities in thyroid stimulating hormone (TSH), free T3 (FT 3), or free T4 (FT4) were not clinically significant as assessed by the investigator, or hypothyroidism was stable under the control of stable hormone replacement therapy.
8. Female patients with fertility must have negative serum pregnancy test during screening, and agree to take effective birth control / contraception to prevent pregnancy from the study period to 6 months after the last administration. Male patients must agree to take effective contraceptive methods from the study period to 6 months after the last administration.

Exclusion Criteria:

1. Have received clinical trial treatment of any other drug or participated in clinical study of medical device within 4 weeks prior to the first drug administration;
2. Prior treatment with immune checkpoint inhibitors (such as pD-1, PD-L1, CTLA-4 and other targeted antibodies) or immune checkpoint agonists (such as ICOS, CD40, CD137, OX40 and other targeted antibodies).
3. Within 4 weeks before the initial administration of the study drug, she had received chemotherapy and radiotherapy (palliative radiotherapy should be completed at least 2 weeks before the initial administration).
4. Have received TCM and/or Proprietary Chinese medicine therapy or immunomodulatory drugs (such as thymosin, interferon, interleukin, etc.) with antitumor effects (according to the instructions) within 2 weeks prior to the first administration of study drugs;
5. Other targeted therapies (such as tyrosine kinase inhibitors) did not exceed 5 half-lives before the first administration;
6. In addition to the tumor that the subject had enrolled in the study, there were other active malignancies within 2 years prior to the first dose. Patients with locally curable tumours (which appear to be cured), such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or carcinoma in situ of the breast, are not excluded.
7. For patients in cohort C:

   A) have pathological types other than squamous carcinoma and adenosquamous carcinoma (e.g., small cell carcinoma, adenocarcinoma, clear cell carcinoma, sarcoma, etc.).

   B) The investigator determined that there was clinically significant hydronephrosis of the renal pelvis or ureter that could not be relieved by nephrostomy or urethral stenting.
8. Before the first administration of the study drug, there were still patients with AE caused by previous antitumor therapy > grade 1 (CTCAE5.0), except for those AE that could not be recovered to ≤ grade 1 as determined by the researcher based on clinical conditions, such as hair loss and fatigue, and which had been in a stable state for a long time;
9. Major surgery (such as craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to initial study drug administration, major surgery is defined here as level 3 or 4; Those with a history of organ transplantation;
10. History of gastrointestinal perforation, gastrointestinal fistula, female genital fistula (such as vesico-vaginal fistula, urethrovaginal fistula, vesico-cervical fistula, etc.) within 6 months before first administration; If the perforation or fistula has been treated, such as removal or repair, and the investigator determines that the disease has recovered or is in remission, enrollment may be permitted.
11. Known to have interstitial lung disease with symptoms that may prevent the discovery or treatment of drug-related pulmonary toxicity during the study.
12. Patients with tumor brain metastases were excluded in the dose escalation phase (asymptomatic patients with brain metastases were allowed in the dose extension phase [asymptomatic duration, i.e. stable condition > 3 weeks, without radiotherapy or glucocorticoid treatment]);
13. Patients who had bleeding from esophageal or gastric varices within the past 6 months, or who were assessed by the investigator to be at risk for bleeding;
14. Serious cardiovascular diseases: New York Heart Association classification (NYHA) is class 2 or above heart failure, left ventricular ejection fraction (LVEF) < 50%, unstable arrhythmia or unstable angina pectoris, uncontrolled hypertension (defined in this protocol as, despite optimal antihypertensive therapy, However, systolic blood pressure > 150mmHg and/or diastolic blood pressure > 100mmHg were clinically significant as assessed by the investigator);
15. Patients with a history of autoimmune diseases (stable hypothyroidism controlled by stable dose thyroid hormone replacement therapy can be included);
16. Patients who are using immunosuppressants, or systemic or absorbable local hormone therapy for immunosuppressive purposes (doses >10mg/ day of prednisone or other equivalent hormone) and continue to use the drug within 2 weeks prior to initial administration of the study drug;
17. The presence of clinically significant active infections requiring intravenous antibiotic treatment, including patients with active tuberculosis;
18. Persons infected with the following diseases: human immunodeficiency virus (HIV) infection; Treponema pallidum antibody positive; Hepatitis B virus infection [hepatitis B surface antigen (HBsAg) or core antibody (HBcAb) positive and HBV DNA test >2000IU/ mL (or 1×104 copies /mL)]; Hepatitis C virus infection [HCV antibody and viral ribonucleic acid (HCV RNA) test positive];
19. Received live/attenuated vaccines within 4 weeks prior to screening or plan to receive live/attenuated vaccines during the study period;
20. Severe hypersensitivity to any monoclonal antibody is known;
21. Patients with a known history of psychotropic substance abuse or drug use that is considered to affect study compliance;
22. Pregnant or lactating women;
23. Other patients considered unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Explore the maximum tolerated dose (MTD) | 21 days after first dosing
  Tolerance evaluation: Dose-limiting toxicity (DLT) is defined as follows: Patients develop the following AE associated with the study drug between day 1 and day 21 after cycle 1 administration: 1)Non-hematological toxicity of grade ≥3 (nausea, vomiting, and diarrhea were relieved within 3 days after supportive treatment, except for infusion reactions that recovered within 2 hours after symptomatic treatment); 2)Grade ≥4 hematologic toxicity (including grade ≥3 neutropenia with fever; However, grade 4 neutropenia requires a duration of ≥7 days to determine DLT); 3) Grade ≥4 thrombocytopenia or grade 3 thrombocytopenia with bleeding.
  Safety evaluation indexes: Safety indicators include: vital signs, physical examination, laboratory tests, electrocardiogram, cardiac color ultrasound, adverse events (including immune-related adverse events), etc.

SECONDARY OUTCOMES:
To evaluate the PK characteristics of BAT1308 injection | 126 days after first dosing
  Blood samples were collected from all dose groups at specific time points during treatment, and 2mL blood samples were collected at each time point to detect the concentration level of BAT1308 in serum and study the pharmacokinetic (PK) characteristics of BAT1308 injection. PK blood samples were collected from subjects before and after each dosing in cycles 1 to 6. In the first and fourth cycles, intensive sampling was carried out to study PK characteristics of steady-state studies of single administration and multiple administration, respectively.
To evaluate the immunogenicity of BAT1308 injection | 126 days after first dosing
  All subjects in the dose groups were required to collect blood samples at specific points during treatment, and 3.5ml blood samples were planned for each time point to detect antidrug antibodies in the serum. For blood samples with positive anti-drug antibodies, further testing of titers and neutralizing antibodies is required.
To evaluate the pharmacodynamics of BAT1308 injection | 126 days after first dosing
  The receptor occupancy of BAT1308 injection was studied by detecting PD-1 receptor binding on T cells in peripheral blood. Subjects in all dose groups required blood samples to be collected at specific points during treatment. Pharmacodynamic receptor occupancy studies were performed only in dose-increasing subjects. 2mL blood samples were collected at each time point, and intensive samples were collected before and at the end of the first cycle, 168h and 336h, respectively, and before the second to sixth cycle.
Preliminary evaluation of the anti-tumor efficacy of BAT1308 injection. | 126 days after first dosing
  The antitumor efficacy of BAT1308 was assessed with RECIST1.1 and iRECIST1.1 throughout the trial. Tumor imaging was performed within 28 days prior to initial dosing, and the same imaging technique was used in the same patient at the same site throughout the study period. If there are brain metastases, do head MRI. RECIST 1.1 was used as the main evaluation criterion. Tumor evaluation after dosing was performed at weeks 6 (D42±5), 12 (D84±5), and 18 (D126±5). The extended study tumor assessment was performed every 9 weeks (±7 days) after week 18 until disease progression, withdrawal of informed consent, loss of follow-up, death, acceptance of new antitumor therapy, or up to 12 months after initial administration, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, M.D, Principal Investigator — Henan Tumor Hospital
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No